CLINICAL TRIAL: NCT00953251
Title: High Sensitive Cardiac Troponin T for Early Prediction of Evolving Non-ST Segment Elevation Myocardial Infarction in Patients With Suspected Acute Coronary Syndrome and Negative Troponin Result on Admission
Brief Title: TnThs Predicting Evolving Non-STEMI
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. med. Evangelos Giannitsis, Department of Cardiology, University of Heidelberg
Other Study IDs: TnT hs 2
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Acute Coronary Syndrome
Keywords: high sensitive troponin T; non-STEMI; early detection.; To detect non-STEMI in a cohort of patients with acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were collected on admission and ideally every hour within the initial 6 hours after admission, unless the patient refused the blood draw, or venipuncture was not feasible due to technical reasons.
  After collection, blood samples were centrifuged immediately and serum stored at -80°C until analysis. The laboratory staff responsible for measurements was blinded to patient data.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with acute coronary syndrome: patients with acute coronary syndrome
- Non-STEMI and unstable angina

SUMMARY:
BACKGROUND: We sought to determine the diagnostic value of the new TnThs assay for early detection of evolving non-STEMI in patients with acute coronary syndrome and a negative 4th generation cTnT result on admission.

METHODS: We evaluated several statistical patterns of blood results of TnT hs and cTnT of 115 patients and calculated necessity of prediction of evolving non-STEMI within 6 hours.

RESULTS: Based on the results of the 4th generation cTnT assay, an evolving non-STEMI was diagnosed in 26 patients, 31 were classified as unstable angina. The TnThs lead to an increase of non-STEMI diagnosis as compared to the 4th generation assay. We could calculate increased sensitivities for earlier detection of evolving non-STEMI from 61.5% on admission to 90.9% within 3 hours and 100% within 6 hours compared to cTnT.

CONCLUSIONS: The TnThs assay enables earlier detection of non-STEMI and allows identification of an additional percentage of cases with non-STEMI previously classified as unstable angina.

ELIGIBILITY:
Inclusion Criteria:

* 115 consecutive patients were enrolled with symptoms suggestive of ACS, admitted to the Chest Pain Unit of the University of Heidelberg. All patients received a 12-lead electrocardiogram (ECG) recording on admission, and a second 12-lead ECG after 6 hours

Exclusion Criteria:

* Patients who underwent percutaneous coronary intervention (PCI) during follow-up sampling were excluded as were patients with a significant kidney dysfunction defined as an estimated glomerular filtration rate below 60 ml/min/1.73m2.
* Patients with STEMI were excluded.
* Patients with only 1 blood sample were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between May 2008 and December 2008, 115 consecutive patients were enrolled with symptoms suggestive of ACS. All patients received a 12-lead electrocardiogram recording on admission, and a second 12-lead ECG after 6 hours. Blood samples were collected on admission and ideally every hour within the initial 6 hours after admission.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to determine the diagnostic accuracy of the new TnThs in subsequent blood draws for earlier detection of evolving non-STEMI in a nonselected population of patients presenting with ischemic symptoms suggestive of ACS. | within 6 hours after admission

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Giannitsis E, Kehayova T, Vafaie M, Katus HA. Combined testing of high-sensitivity troponin T and copeptin on presentation at prespecified cutoffs improves rapid rule-out of non-ST-segment elevation myocardial infarction. Clin Chem. 2011 Oct;57(10):1452-5. doi: 10.1373/clinchem.2010.161265. Epub 2011 Aug 1. PMID 21807867